CLINICAL TRIAL: NCT04967027
Title: Safety and Tolerability of TTFields for Patients With Brain Metastases After the Standard Treatment Fails: a Prospective, Single-center, Single-arm Study
Brief Title: Phase 1 Trial for Tumor Treating Field for Drug/Radiation Resistant Brain Metastases
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: BM V1.0/2020-08-01
Record Dates: First submitted 2021-07-04; First posted 2021-07-19 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-07

CONDITIONS: Brain Metastases
Keywords: Tumor Treating Fields; Brain metastases;
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TTFields group (Experimental): patients with brain metastases who have been resistant to drug or radiation therapy, to be treated by continuous TTFields treatment using the ASCLU-300 TTF device.
  Interventions: Device: ASCLU-300 TTF

INTERVENTIONS:
Device: ASCLU-300 TTF — BM treated by continuous TTFields treatment (ASCLU-300, approved by Chinese FDA)

SUMMARY:
Brain metastasis is a very common disease with poor prognosis, 20% cancer will develop brain metastases(BM), up to 40% by autopsy. Great advances have made with the application of targeting therapy, immunotherapy, chemotherapy, whole brain radiation and radiosurgery, however, treated patients were finally suffered from drug/radiation resistance and rapid recurrence. Tumor treating fields (TTFields) is one of the standard combination treatment for GBM, and some researchers believe that TTFields can effectively inhibit patient-derived lung adenocarcinoma brain metastasis cells progression in vitro. In this study, the investigator attempts to evaluate the safety, and tolerability of TTFields in adult participants diagnosed with Drug/Radiation resistant BM.

ELIGIBILITY:
Inclusion Criteria:

* patients are diagnosed as brain metastases by Xiangya Hospital multidisciplinary team;
* age from 18 to 65 year-old;
* patients have been progressed from standard therapy (drug/radiation resistance)
* KPS more than 70 score;
* anticipated OS more than 3 months;
* signed consent form.

Exclusion Criteria:

* unable to take TTFields more than 18 hours each day;
* unable to follow-up till progression;
* the scalp wound is not well healed, the head skin condition is not good, the skull has a large area defect, or other situations that are not suitable for wearing electrodes
* pregnant women;
* last drug within 4 weeks, last radiation within 3 months, take other trials;
* other heavy diseases like heavy infection;
* other condition: Such as breastfeeding, installation of cardiac pacemakers, brain stimulators, severe intracranial edema, increased intracranial pressure leading to midline structures exceeding 5 mm, optic nerve head edema, disturbance of consciousness, etc., allergies to conductive coupling agents, gels, etc.
* blood and biochemical indicators in the following range: A. Liver function impairment: AST or ALT > 3 times the upper limit of normal; B. Total bilirubin> upper limit of normal value; C. Renal impairment: serum creatinine>1.7mg /dL (>150 mol/L); D. Coagulopathy: PT or APTT >1.5 times normal; E. Platelets counts < 100x10^9/L; F. Absolute neutrophils count < 1x10^9/L; G. Hemoglobin < 100g/L;
* other conditions physicians not suggest to take the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The treatment-related adverse events | 12 months
  Number of patients who experienced a treatment-related adverse event.
Time to Progression | 12 months
  Time to progression of patients with brain metastases
Overall Survival Rate | 12 months
  Number of patients alive at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiong Liu, MD, Principal Investigator — Xiangya Hospital of Central South University; Yu Zeng, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided
due to protect the patients' privacy, we have not yet decided to share each IPD, but we can share IPD once other researchers request upon approval by our Ethics Committee